CLINICAL TRIAL: NCT04887883
Title: Influence of Sex, Acute Resistance Exercise and Training on de Novo Muscle Protein Synthesis
Brief Title: Influence of Sex and Training on de Novo Muscle Protein Synthesis
Acronym: TUT
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Daniel Moore, Professor, University of Toronto
Other Study IDs: TUT study; RGPIN-2015-04521 (Other Grant/Funding Number: NSERC Discovery Grant)
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Amino Acids; Dietary Protein; Sex; Resistance Exercise
Keywords: intrinsically labeled proteins; muscle protein synthesis
MeSH Terms: conditions — Coitus | interventions — Resistance Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Muscle biopsies, blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males: 10 young healthy biological males aged 18 - 30 y
  Interventions: Behavioral: Resistance exercise
- Females: 10 young healthy biological females aged 18 - 30 y
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — Participants performed 8 weeks of resistance training and muscle biopsies were taken before and 24 h before and after the program.

SUMMARY:
Acute exercise increases the incorporation of dietary amino acids into de novo myofibrillar proteins after a single meal in controlled laboratory studies in males. It is unclear if this extends to free-living settings or is influenced by training or sex. Over 24 h in a free-living setting, the investigators determined the effect of training status and sex on dietary phenylalanine incorporation into contractile myofibrillar and noncontractile sarcoplasmic proteins after exercise.

DETAILED DESCRIPTION:
Exogenous (e.g. diet-derived) amino acids increase muscle protein synthesis and provide the building blocks for growth. While traditional infusion studies can measure the synthesis of total mixed muscle or fraction-specific protein synthetic rates, the metabolic fate of dietary amino acids can only be assessed by measuring the incorporation of a labelled amino acid (i.e. L-[1-13C]phenylalanine) into muscle protein through the oral ingestion of a intrinsically labelled food source (e.g. milk protein) . This technique has revealed in controlled laboratory settings that dietary amino acids, and not endogenous amino acids recycled from intracellular protein breakdown, may be preferentially utilized as precursors for muscle and whole body protein synthesis Therefore, it is important to characterize the incorporation of diet-derived amino acids over a 24-h post-exercise recovery period to determine how RE influences their utilization as precursors for the synthesis of new muscle proteins. The investigators are unaware of any studies that have examined the utilization of dietary amino acids for de novo muscle protein synthesis in females, highlighting an urgent need to rectify the sex-disparity in exercise-related research.

Protein requirements during resistance training have been suggested to be highest at training onset with evidence suggesting moderate daily intakes (~1.2-1.4 g·kg·d-1) can support chronic adaptations, although recent suggestions are that slightly higher intakes (~1.6 g·kg·d-1) may optimize lean mass growth. Resistance training is associated with a reduction in whole-body protein turnover but an increased net protein balance suggesting a greater efficiency of whole-body amino acid utilization with training in males , although whether this also extends to females is unknown. Acute RE and chronic training has been reported to increase intracellular amino acid recycling in the fasted state, which would be consistent with an increased amino acid efficiency. To date, however, no study has investigated whether the post-exercise incorporation of dietary amino acids into myofibrillar and sarcoplasmic proteins in a free-living setting is modified by training and/or sex.

The primary aim of the present study was to determine the dietary fate of amino acids into contractile myofibrillar and noncontractile sarcoplasmic muscle proteins after acute RE in the untrained and trained state over 24 h in a free-living setting. The investigators hypothesized that, irrespective of sex, acute RE would increase dietary amino acid incorporation in myofibrillar proteins in the untrained state with training leading to an attenuated increase suggestive of a reduced reliance on dietary amino acids in the trained state.

ELIGIBILITY:
Inclusion Criteria:

* Participants were included in the study after reporting not engaging in whole body RE or plyometrics in the past 3 months and had a BMI between 18.5-27.5 kg/m2.
* Females were included if they had a regular menstrual cycle with the last 3 months and

Exclusion Criteria:

* Participants were excluded if they: i) consumed tobacco and/or illicit anabolic drug use (e.g. testosterone, growth hormones); ii) were a vegan or had a nut allergy and; iii) participated in a study within the past year involving stable isotopes.
* Females were excluded if they used oral contraceptives and/or discontinued their use within the last 3 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: : Ten recreationally active and healthy young males and females
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Dietary fate of amino acids into myofibrillar and sarcoplasmic proteins | The change in muscle MPE at 0 and 24 h after acute resistance exercise before and after training
  MPE

SECONDARY OUTCOMES:
Amino acid transporter protein content | 0 and 24 hours after acute resistance exercise before and after training
  Arbitrary units
mTOR localization with capillaries | 0 and 24 hours after acute resistance exercise before and after training
  Pearson's r

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abou Sawan S, Hodson N, Malowany JM, West DWD, Tinline-Goodfellow C, Brook MS, Smith K, Atherton PJ, Kumbhare D, Moore DR. Trained Integrated Postexercise Myofibrillar Protein Synthesis Rates Correlate with Hypertrophy in Young Males and Females. Med Sci Sports Exerc. 2022 Jun 1;54(6):953-964. doi: 10.1249/MSS.0000000000002878. Epub 2022 Jan 25. PMID 35081094